CLINICAL TRIAL: NCT04902638
Title: Continuous Glucose Monitoring in Total Knee Arthroplasty With Preoperative High Dose Dexamethasone: A Randomized Controlled Study
Brief Title: Continuous Glucose Monitoring in Total Knee Arthroplasty With Preoperative High Dose Dexamethasone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Glucose Monitor TKR
Record Dates: First submitted 2021-05-20; First posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Diabetes; Knee Osteoarthritis
MeSH Terms: conditions — Diabetes Mellitus; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Diabetic patients with steroid (Active Comparator)
  Interventions: Procedure: Intraarticular injection of dexamethasone
- Diabetic patients without steroid (Placebo Comparator): Injection of normal saline
  Interventions: Procedure: Intraarticular injection of dexamethasone
- Pre-diabetic patients with steroid (Active Comparator)
  Interventions: Procedure: Intraarticular injection of dexamethasone
- Pre-diabetic patients without steroid (Placebo Comparator): Injection of normal saline
  Interventions: Procedure: Intraarticular injection of dexamethasone
- Non-diabetic patients with steroid (Active Comparator)
  Interventions: Procedure: Intraarticular injection of dexamethasone
- Non-diabetic patients without steroid (Placebo Comparator): Injection of normal saline
  Interventions: Procedure: Intraarticular injection of dexamethasone

INTERVENTIONS:
Procedure: Intraarticular injection of dexamethasone — Intraarticular injection of dexamethasone

SUMMARY:
Perioperative joint infection (PJI) is a rare but serious postoperative complication from total knee arthroplasty (TKA) and it is known to cause significant morbidities to the patients suffering from it. Literatures have found evidence that there is correlation between patients' perioperative blood glucose level and their risks of developing PJI postoperatively. By monitoring patients' perioperative blood glucose level, clinicians may be able to better identify patients who are at risks of developing PJI.

Continuous blood glucose level monitoring, where patients carry a blood glucose monitoring device, has been a novel intervention in various medical specialties for recording and monitoring patients' blood glucose levels. However, currently there has only limited studies using this intervention for perioperative blood glucose monitoring in patients who are receiving total knee arthroplasty.

Intravenous dexamethasone is a widely used treatment for patients undergoing total knee arthroplasty as it has been shown in previous studies that it can provide good analgesic effect and also reduce patients' nauesea symptoms preoperatively. However, hyperglycaemia is also a known side effects from dexamethasone. There still has not been ample amount of investigation on how significant this potential effect is and at what period of time perioperatively that this side effect occurs.

This study is designed to investigate how intravenous dexamethasone can potentially affect the perioperative blood glucose levels in patients receiving total knee arthroplasty. And by using a continuous glucose monitoring machine we are also aiming to find out the variability of the perioperative blood glucose profiles of these patients in order to design a better glucose monitoring schedule.

DETAILED DESCRIPTION:
Perioperative joint infection (PJI) is a rare but serious postoperative complication from total knee arthroplasty (TKA) and it is known to cause significant morbidities to the patients suffering from it. Literatures have found evidence that there is correlation between patients' perioperative blood glucose level and their risks of developing PJI postoperatively. By monitoring patients' perioperative blood glucose level, clinicians may be able to better identify patients who are at risks of developing PJI.

Continuous blood glucose level monitoring, where patients carry a blood glucose monitoring device, has been a novel intervention in various medical specialties for recording and monitoring patients' blood glucose levels. However, currently there has only limited studies using this intervention for perioperative blood glucose monitoring in patients who are receiving total knee arthroplasty.

Intravenous dexamethasone is a widely used treatment for patients undergoing total knee arthroplasty as it has been shown in previous studies that it can provide good analgesic effect and also reduce patients' nauesea symptoms preoperatively. However, hyperglycaemia is also a known side effects from dexamethasone. There still has not been ample amount of investigation on how significant this potential effect is and at what period of time perioperatively that this side effect occurs.

This study is designed to investigate how intravenous dexamethasone can potentially affect the perioperative blood glucose levels in patients receiving total knee arthroplasty. And by using a continuous glucose monitoring machine we are also aiming to find out the variability of the perioperative blood glucose profiles of these patients in order to design a better glucose monitoring schedule.

ELIGIBILITY:
Inclusion Criteria:

* Obtained informed consent
* Adult patients (>18 years old)
* Primary osteoarthritis of knees scheduled for unilateral TKA

Exclusion Criteria:

* Unable to obtain consent
* Refusal to continuous glucose monitoring
* Contraindication to dexamethasone
* Patients scheduled for one-staged bilateral Total Knee Arthroplasty (TKA)
* History of peptic ulcer/GI bleeding
* Hepatitis B carrier
* Patients on long-term steroid
* Patients requiring general anesthesia for the operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Hyperglycaemia time | Within 1 week of admission
  Amount of time where patients are at hyperglycaemic state

CONTACTS AND LOCATIONS:
Overall Officials: Lik Hang Brian Leung, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- Duchess of Kent Children Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No